CLINICAL TRIAL: NCT02398630
Title: "Estudio de Histerosalpingografía Por Resonancia Magnética Para la evaluación Integral de la Paciente infértil."
Brief Title: "Magnetic Resonance Imaging Hysterosalpingography for the Integral Evaluation of the Infertile Patient."
Acronym: HSG-RM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diagnostico Maipu (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSG-RM
Record Dates: First submitted 2015-03-20; First posted 2015-03-25 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Women Infertility
Keywords: Histerosalpingography; MRI; Magnetic Resonance Imaging; HSG; Diagnostico Maipu; Imaging; Carrascosa Patricia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label (Other): This is a single arm open label study.
  Its procedures involve:
  * Transvaginal Echography
  * Conventional Virtual Histerosalpingography
  * Virtual Histerosalpingography by MRI
  * Blood draw for Antimullerian Hormone Dosing
  Interventions: Radiation: TC Virtual Hysterosalpingography; Other: MRI Virtual Hysterosalpingography; Other: Antimullerian Hormone dosing; Other: Transvaginal Echography

INTERVENTIONS:
Radiation: TC Virtual Hysterosalpingography — Virtual hysterosalpingography: a new multidetector CT technique for evaluating the female reproductive system
  Other Names: HSG-V
Other: MRI Virtual Hysterosalpingography — Magnetic Resonance Imaging Virtual hysterosalpingography
  Other Names: HSG-MRI
Other: Antimullerian Hormone dosing — Blood Draw for Antimullerian Hormone dosing
Other: Transvaginal Echography — Transvaginal Echography for evaluating the female reproductive system
  Other Names: TV-Echo

SUMMARY:
Abstract:

Recent advances in reproductive medicine have generated a demand for more accurate imaging methods for identifying the specific cause of female infertility and other gynecologic disorders. Virtual hysterosalpingography is an emerging modality in which aspects of the established technique of hysterosalpingography are combined with the cutting-edge technology of multidetector computed tomography (CT) to allow a comprehensive and highly accurate evaluation of both the female reproductive system and the pelvic anatomy generally. Unlike ultrasonography (US) and magnetic resonance (MR) imaging, multidetector CT is capable of depicting both the external and internal surfaces of the uterus, fallopian tubes, and other pelvic organs, providing high-resolution data that are suitable for two- and three-dimensional reconstructions and virtual endoscopic views. Thus, virtual hysterosalpingography may prove to be superior to other noninvasive modalities for evaluating tubal patency. Moreover, in comparison with conventional hysterosalpingography, which may involve cervical clamping, virtual hysterosalpingography is painless. Because of the health risks associated with ionizing radiation, the use of another modality (eg, MR imaging, US) may be preferred if the presence of a focal uterine lesion is strongly suspected. However, virtual hysterosalpingography with multidetector CT may provide a diagnostic advantage in complex cases.

DETAILED DESCRIPTION:
Infertility is a common problem that affects one in six couples. It is defined as the inability to get pregnant after a reasonable time (12 months) of sex without using birth control measures. The causes of the increased prevalence of infertility are difficult to establish. This increase could be due to several factors such as the postponement of the time when it is decided to have children, alterations in semen quality, changes in sexual behavior, etc. The study of the infertile couple has always been focussed on different factors: ovulatory (20%), utero-tubal (30%) , the migration of sperm (10%) and male (30%). About 40% of all infertile couples exhibit a combination of factors and about 15% do not display any objective alteration leading to a definite diagnosis.

During the last two decades major changes occurred in the approach to infertility. With the introduction of new assisted reproductive technologies, the development of molecular biology and novel diagnostic imaging methods, there have been major advances in the evaluation and treatment of couples considered infertile.

Hysterosalpingography (HSG) is the useful imaging method for evaluating the fallopian tubes and uterine cavity. Scanning is performed in the follicular phase of the cycle and is carried out in an X-ray fluoroscopy. Indications for HSG have been reduced with the introduction of new diagnostic methods, actually being basically an essencial technique used in the study of the factors responsible for infertility as well as recurrent abortions. On the downside, exposure to radiation and use of impingement of the cervix during the procedure, with the possible complications mentioned.

Due to technological advances, a new technique based on CT studies has been developed, and it is called virtual Hysterosalpingography (HSG-V). It is performed with a multislice CT scanner with high resolution and quality of images. It is a noninvasive study and needs none pinch the cervix. It has the ability to assess blockages and defects or other uterine and tubal problems, besides appreciating for abnormalities that may cause the inability of a couple to achieve pregnancy. Also reveals the organs of the pelvis in its entirety and fallopian tubes, and inside its walls. This helps to detect the presence of polyps, adhesions, fibroids, narrow tubes, or occupying lesions light. Compared with conventional HSG, the advantage is that it is non-invasive, painless and takes only a few seconds, conditions that provide women with greater comfort. Moreover, it provides the doctor with more complete information than the conventional method, because it provides two-dimensional and three-dimensional endoscopic images. Additionally, the radiation received by the patient is less than that required in the conventional study.

Magnetic resonance imaging (MRI) of the female pelvis is the largest study performance evaluation of pelvic pathology (endometriosis, fibroids, adenomyosis, etc.). Contributing to this characteristics of being non-invasive and does not use ionizing radiation. It has high resolving power for the assessment of ovarian and uterine pathology, being especially useful for cases where ultrasound is inconclusive. It also plays a dual role in the case of uterine malformations: It allows the extension and/or confirmation of the ultrasound diagnosis and evaluates the associated malformations, mainly of the urinary system. Major limitations of the MRI are low availability, presence of a pacemaker or metallic foreign bodies. A relative advantage is its lower cost compared to the HSG-V, and lower cost if making multiple conventional studies.

Current assessment of the patient with infertility involves several studies to determine the causative factor. The virtues of the MRI position it as an integrative alternative to conventional multi-modal methods in the study of the female pelvis.

ELIGIBILITY:
Inclusion Criteria:

* Requested Virtual Hysterosalpingography.
* Diagnosis of Infertility.
* Informed Consent.

Exclusion Criteria:

* Pregnancy at the time of examination.
* Carriers of pacemaker devices.
* Ferromagnetic elements incompatible with MRI.
* Claustrophobia.
* Allergy to iodine.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Tubal patency | Six months
  Evaluation of the tubal patency between CT and MRI
Endocavitary pathology | Six months
  Evaluation of endocavitary pathology between US, CT and MRI

SECONDARY OUTCOMES:
Antral follicle count | Six months
  Comparison of antral follicle count between US and MRI and its correlation with antimullerian hormone

CONTACTS AND LOCATIONS:
Locations (1):
- Diagnostico Maipu, Vicente López, Buenos Aires, Argentina

REFERENCES:
- See also: Diagnostico Maipu Website — http://www.diagnosticomaipu.com